CLINICAL TRIAL: NCT01208441
Title: A Phase Ib Neoadjuvant Study of the Gamma Secretase Inhibitor (RO4929097) in Combination With the Aromatase Inhibitor Letrozole in Post-Menopausal Women With Stage II/III Hormone Receptor-Positive Breast Cancer
Brief Title: RO4929097 and Letrozole in Treating Post-Menopausal Women With Hormone Receptor-Positive Stage II or Stage III Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02487; NCI-2011-02487 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UPCI-09-080; CDR0000683397; UPCI 09-080 (Other: University of Pittsburgh Cancer Institute); 8554 (Other: CTEP); U01CA099168 (NIH)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Arm I (Experimental): Patients receive oral letrozole once daily on days 1-21. Beginning in course 2, patients also receive oral RO4929097 on days 1-3, 8-10, and 15-18. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Beginning 1 week after completion of neoadjuvant therapy, patients undergo surgery or tumor biopsy. Patients continue to receive oral letrozole once daily during surgery and for an additional 4 weeks.
  Interventions: Drug: letrozole; Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Procedure: therapeutic conventional surgery; Procedure: breast biopsy; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: letrozole
  Other Names: CGS 20267; Femara; LTZ
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097
  Other Names: R4733; RO4929097
Procedure: therapeutic conventional surgery
Procedure: breast biopsy
  Other Names: biopsy of breast
Other: diagnostic laboratory biomarker analysis
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of RO4929097 when given together with letrozole in treating post-menopausal women with stage II or stage III breast cancer. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving RO4929097 together with letrozole may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum-tolerated dose and the recommended phase II dose of gamma-secretase inhibitor RO4929097 (RO4929097) in combination with letrozole in post-menopausal women with hormone receptor-positive stage II or III breast cancer.

II. To assess the safety of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of this regimen, taking into consideration the induction of CYP3A4, in these patients.

II. To characterize the pharmacodynamic effects of letrozole prior to and during administration of RO4929097 with attention to suppression of estradiol and estrone levels.

III. To describe the pharmacodynamic effects of letrozole with or without RO4929097 on the NOTCH pathway, proliferation, angiogenesis, stromal cell infiltration/pathways, and comprehensive genomic analysis in tumor tissue of these patients.

IV. To describe the response, including clinical complete or partial objective response, pathological complete response, and attainment of pathologic stage 0 or I status in these patients.

OUTLINE: This is a multicenter, dose-escalation study of gamma-secretase inhibitor RO4929097(RO4929097).

Patients receive oral letrozole once daily on days 1-21. Beginning in course 2, patients also receive oral RO4929097 on days 1-3, 8-10, and 15-18. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Beginning 1 week after completion of neoadjuvant therapy, patients undergo surgery or tumor biopsy. Patients continue to receive oral letrozole once daily during surgery and for an additional 4 weeks.

Blood and tumor tissue samples are collected at baseline and periodically during study for pharmacokinetics, pharmacodynamics, and correlative studies.

After completion of study therapy, patients are followed up for 1 month and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast cancer

  * Stage II or III disease (T2-T3, N0-2)

    * No N3, T4 disease
  * Estrogen receptor-positive (ER+) and/or progesterone receptor-positive (PR+)

    * H score ≥ 10 or positivity ≥ 10%
  * HER2 negative as determined by IHC (1 or 2+) or FISH (< 2.0+)
* Bilateral disease allowed as long as all tumors are ER+ and ≥ 1 is T2-T3
* Patient must have disease that is palpable on physical exam and able to be imaged via breast ultrasound

  * Defined as ≥ 1 T2 tumor > 2 cm
  * Multifocal disease allowed provided that ≥ 1 of the tumors is > 2 cm
* No metastatic disease by CT scans of the chest, abdomen, and pelvis, a PET/CT bone scan, or nuclear medicine bone scan
* No inflammatory breast cancer or presence of breast tumor cells in the dermal lymphatics of the breast
* Post-menopausal meeting 1 of the following criteria:

  * Bilateral oophorectomy
  * Age ≥ 50 years and amenorrheic for > 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression (spontaneous amenorrhea)
* ECOG performance status (PS) 0-2 (Karnofsky PS 60-100%)
* Life expectancy > 3 months
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Baseline QTcF ≤ 470 msec
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma secretase inhibitor RO4929097 or other agents used in the study
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* Able to swallow tablets
* Not serologically positive for hepatitis A, B, or C, or have a history of liver disease, other forms of hepatitis, or cirrhosis
* No uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia despite adequate electrolyte supplementation
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * History of torsades de pointes or other significant cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* Recovered to < grade 2 CTCAE toxicities related to prior therapy
* No prior chemotherapy, hormonal therapy, radiotherapy, or biological therapy for breast cancer

  * Prior treatment for non-melanoma skin cancer or carcinoma in situ of the cervix allowed
  * No prior hormone therapy for ductal carcinoma in situ (DCIS)
* No other concurrent investigational agents
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers and/or inhibitors or substrates of CYP3A4

  * Switching to alternative medications allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent antiarrhythmics or other medications known to prolong QTc
* No other concurrent anticancer agents or therapies
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level at which no more than 1 of 6 patients experience a DLT, and the dose below that at which at least 2/6 patients have DLT according to NCI CTCAE version 4.0 | 21 days

SECONDARY OUTCOMES:
Measurement of NOTCH 1 and 4, activated NOTCH (ICN), Hey 1 and NOTCH ligands (DLL4 and Jagged 1) | Baseline
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of NOTCH 1 and 4, activated NOTCH (ICN), Hey 1 and NOTCH ligands (DLL4 and Jagged 1) | 21 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of NOTCH 1 and 4, activated NOTCH (ICN), Hey 1 and NOTCH ligands (DLL4 and Jagged 1) | 42 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of NOTCH 1 and 4, activated NOTCH (ICN), Hey 1 and NOTCH ligands (DLL4 and Jagged 1) | At time of surgery
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Genomic analysis of RNA transcriptome, mirco-RNA transcriptome, and DNA methylation | Baseline
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value. For the analysis of the gene expression data, the overall false discovery rate (FDR), which is defined as the expected portion of false positives, will be controlled at 20% to generate a list of genes for further investigation.
Genomic analysis of RNA transcriptome, mirco-RNA transcriptome, and DNA methylation | 21 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value. For the analysis of the gene expression data, the overall FDR, which is defined as the expected portion of false positives, will be controlled at 20% to generate a list of genes for further investigation.
Genomic analysis of RNA transcriptome, mirco-RNA transcriptome, and DNA methylation | 42 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value. For the analysis of the gene expression data, the overall FDR, which is defined as the expected portion of false positives, will be controlled at 20% to generate a list of genes for further investigation.
Genomic analysis of RNA transcriptome, mirco-RNA transcriptome, and DNA methylation | At time of surgery
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value. For the analysis of the gene expression data, the overall FDR, which is defined as the expected portion of false positives, will be controlled at 20% to generate a list of genes for further investigation.
Measurement of cell proliferation (Ki-67) | Baseline
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of cell proliferation (Ki-67) | 21 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of cell proliferation (Ki-67) | 42 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of cell proliferation (Ki-67) | At time of surgery
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of appoptosis (TUNEL and activated caspase) | Baseline
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of appoptosis (TUNEL and activated caspase) | 21 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of appoptosis (TUNEL and activated caspase) | 42 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of appoptosis (TUNEL and activated caspase) | At time of surgery
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of angiogenesis (VEGF and CD31) | Baseline
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of angiogenesis (VEGF and CD31) | 21 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of angiogenesis (VEGF and CD31) | 42 days
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.
Measurement of angiogenesis (VEGF and CD31) | At time of surgery
  All measurements are continuous. Descriptive statistics will be calculated to summarize change of each measurement from the baseline value. A two-sided Wilcoxon signed rank test will be used to compare each measurement at a specific time to the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Puhalla, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania